CLINICAL TRIAL: NCT03159975
Title: A Open-label, Dose Escalation, Phase 1 Clinical Trial to Evaluate the Tolerability, Safety and Immunogenicity of GX-70, a DNA-based Therapeutic Vaccine, Administered Intramuscularly by Electroporation (EP) in Patients With Pulmonary Tuberculosis Who Have High Risk Factors for Relapse or Treatment Failure
Brief Title: Safety and Immunogenicity Study of GX-70 in TB Patient
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unconfirmed research expenses
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2016-1144
Record Dates: First submitted 2017-05-14; First posted 2017-05-19 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Tuberculoses; High Risk Factors for Relapse; Treatment Failure
Keywords: Tuberculosis; DNA vaccine; Electroporation; GX-70
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Intervention Model Description: 1. Dose level 1 : GX-70 0.26mg
  2. Dose level 2 : GX-70 1mg
  3. Dose level 3 : GX-70 4mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (GX-70 0.26mg) (Experimental): Administrating GX-70 0.26mg
  Interventions: Drug: GX-70 by electroporation
- Dose level 2 (GX-70 1mg) (Experimental): Administrating GX-70 1mg
  Interventions: Drug: GX-70 by electroporation
- Dose level 3 (GX-70 4mg) (Experimental): Administrating GX-70 4mg
  Interventions: Drug: GX-70 by electroporation

INTERVENTIONS:
Drug: GX-70 by electroporation — Gx-70 0.26mg will be administered by electroporation in the deltoid muscles every 4 weeks 5 times
  Arms: Dose level 1 (GX-70 0.26mg)
Drug: GX-70 by electroporation — Gx-70 1mg will be administered by electroporation in the deltoid muscles every 4 weeks 5 times
  Arms: Dose level 2 (GX-70 1mg)
Drug: GX-70 by electroporation — Gx-70 4mg will be administered by electroporation in the deltoid muscles every 4 weeks 5 times
  Arms: Dose level 3 (GX-70 4mg)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immunogenicity in patients with pulmonary tuberculosis of an investigational DNA vaccine being developed for the prevention of relapse of tuberculosis.

DETAILED DESCRIPTION:
Tuberculosis still matters in domestic as well as global public health. According to WHO, 8,700,000 cases of tuberculosis occured in 2011, and 1,400,000 of them resulted dead. Tuberculosis patients with the cavity and positive on AFB show high rate of relapse and treatment failure. Those with high risk of relapse and treatment failure may need more effective treatment before acquiring resistance and infecting others. GX-70, which consists of the four-antigen plasmids from MTB together with recombinant Flt3 ligand is an investigational DNA vaccine designed to prevent relapse or treatment failure.

The purpose of this study is to assess safety of GX-70, in pulmonary TB patients with high risk factors for treatment failure or relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily consented, after listening enough explanation for this study and investigational product.
2. Adults between 19 and 65 years.
3. TB patients without a history of TB diagnosis, who show positive on both AFB smear and TB-PCR
4. TB patients who satisfy following conditions: cavity spotted from chest imaging before TB therapy, positive on AFB smear 2 months after TB therapy.

Exclusion Criteria:

1. At 2 months after therapy started, AFB smear shows 1+ or higher, but TB PCR shows NTM positive.
2. If positive on AFB smear is resulted from dead MTB
3. Serious TB such as tuberculous encephalomeningitis
4. Patients with serious pulmonary symptom except TB
5. Patients show poor vital sign considered to be difficult to participate
6. Patients with heart, renal, or liver failure
7. Patients with infection, ulcer, edema, tattoo, scar, wound and other conditions in skin around 3cm of deltoid muscle that result inappropriate to inject through electroporation.
8. When thickness of skin around deltoid muscle which is to be injected exceeds 40mm
9. Patients with QTc prolongation on 12-lead ECG
10. Patients with a cardiac device (such as a pacemaker)
11. Patients that the researchers do not think fit into the group, including patients failed in compliance assessment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ability to avoid pregnancy during the trial: Women physically capable of pregnancy must avoid pregnancy during ongoing period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), or use of acceptable contraception: hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD).
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
MTD (Maximum Tolerant Dose) | Every 4 weeks up to 16 weeks

SECONDARY OUTCOMES:
IFN-γ (SFC/106 cells) | Every 8 weeks up to 24 weeks
  IFN-γ response stimulated by TB antigens
Flt3L concentration (pg/ml) | Every 8 weeks up to 24 weeks
  Every 8 weeks up to 24 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flynn JL, Chan J. Tuberculosis: latency and reactivation. Infect Immun. 2001 Jul;69(7):4195-201. doi: 10.1128/IAI.69.7.4195-4201.2001. No abstract available. PMID 11401954
- [Result] Chang KC, Leung CC, Yew WW, Ho SC, Tam CM. A nested case-control study on treatment-related risk factors for early relapse of tuberculosis. Am J Respir Crit Care Med. 2004 Nov 15;170(10):1124-30. doi: 10.1164/rccm.200407-905OC. Epub 2004 Sep 16. PMID 15374844
- [Result] Ahn SS, Jeon BY, Kim KS, Kwack JY, Lee EG, Park KS, Sung YC, Cho SN. Mtb32 is a promising tuberculosis antigen for DNA vaccination in pre- and post-exposure mouse models. Gene Ther. 2012 May;19(5):570-5. doi: 10.1038/gt.2011.140. Epub 2011 Sep 29. PMID 21956689